CLINICAL TRIAL: NCT01764698
Title: Adaptation of CALM for Comorbid Anxiety and Substance Use Disorders
Brief Title: Delivery of Anxiety Disorder Treatment in Addictions Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kate Taylor, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7K23DA031677 (NIH)
Record Dates: First submitted 2012-12-17; First posted 2013-01-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Anxiety Disorders; Substance Use Disorders
Keywords: anxiety disorders; substance use disorders; treatment effectiveness; cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CALM-SUD (Experimental): Participants receive the adaptation of the Coordinated Anxiety Learning and Management (CALM) protocol that demonstrated effectiveness in a large primary care sample. CALM will be adapted for those with anxiety and substance use disorder comorbidity, and will consist of an orientation session and 6 group treatment sessions. These participants will also receive substance abuse treatment as usual at a community Intensive Outpatient Program.
  Interventions: Behavioral: CALM-SUD
- Treatment as usual (Active Comparator): Participants in this arm receive the standard Intensive Outpatient treatment for their substance use disorder at a community addictions treatment facility.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: CALM-SUD — 6-session group for anxiety disorders. Cognitive behavioral therapy including self-monitoring, relaxation, cognitive restructuring, exposure therapy, and relapse prevention. In addition, participants in this arm are also enrolled in an Intensive Outpatient Program for their substance use disorder. The program is run by an outpatient addictions facility and includes up to 16 weeks of groups that meet 3 to 4 times per week in addition to up to 10 individual sessions of therapy. The group model includes motivational interviewing, cognitive behavioral therapy, contingency management, and relapse prevention skills.
  Arms: CALM-SUD
Behavioral: Treatment as usual — The program is run by an outpatient addictions facility and includes up to 16 weeks of groups that meet 3 to 4 times per week in addition to up to 10 individual sessions of therapy. The group model includes motivational interviewing, cognitive behavioral therapy, contingency management, and relapse prevention skills.
  Arms: Treatment as usual

SUMMARY:
Anxiety disorders are highly prevalent among those with substance use disorders, but the majority of addictions treatment centers provide little to no evidence-based treatment for anxiety disorders. Furthermore, tension reduction models suggest that treating anxiety should also improve substance use outcomes. This study is aimed at improving symptoms for people who have substance use and anxiety problems. The study is comparing regular Intensive Outpatient treatment for addiction to Intensive Outpatient treatment for addiction plus treatment for anxiety disorders. Clinicians at a community addictions clinic will participate by receiving training in delivering cognitive behavioral therapy for anxiety disorders and will deliver the treatment to the patient participants. They will also complete some questionnaires. Patient participants will be asked to complete a baseline assessment. Those who are eligible will be randomly assigned to one of the two treatment groups. Those who are assigned to addiction treatment as usual will continue their regular care at the Matrix Institute. Participants who are assigned to also receive the anxiety treatment will be asked to participate in 6, 90-min treatment sessions and an orientation session. All participants will be asked to complete post-treatment and follow-up assessments. The assessments should take approximately 1 hour, and the follow-up assessment will be completed 6 months after treatment is over. It is hypothesized that those who get the additional anxiety disorder treatment will show greater improvement in anxiety and substance use outcomes than those who get Intensive Outpatient Program without the anxiety disorder treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* speak English
* meet diagnostic criteria for at least one anxiety disorder
* score at least an 8 on the OASIS (see Assessments), indicating at least moderate but clinically significant anxiety symptoms
* be enrolled in the Intensive Outpatient Program (IOP) at the Matrix Institute (community partner)
* meet diagnostic criteria for substance abuse or dependence

Exclusion Criteria:

* have unstable medical conditions
* marked cognitive impairment
* active suicidal intent or plan
* active psychosis
* unstable Bipolar I disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Brief Symptom Inventory | baseline, 6 weeks, 6 months
  Change over time is being assessed.
Timeline Follow Back | baseline, 6 week, 6 month
  Change over time is being assessed
Overall Anxiety Severity and Impairment Scale | baseline, 6 week, 6 month
  Change over time is being assessed.

SECONDARY OUTCOMES:
urine toxicology screen | baseline, 6 week, 6 month
  Change over time is being assessed.
Patient Health Questionnaire-8 | baseline, 6 week, 6 month
  brief depression measure; Change over time is being assessed.
Anxiety Sensitivity Index | baseline, 6 week, 6 month
  Change over time is being assessed.
Panic Disorder Severity Scale | baseline, 6 week, 6 month
  Change over time is being assessed.
Social Phobia Inventory | baseline, 6 week, 6 month
  Change over time is being assessed.
Penn State Worry Questionnaire | baseline, 6 week, 6 month
  Change over time is being assessed.
Posttraumatic Stress Disorder Checklist | baseline, 6 week, 6 month
  Change over time is being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kate B Taylor, Ph.D., Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Matrix Institute on Addictions, Los Angeles, California
  - University of California-Los Angeles, Department of Psychiatry and Biobehavioral Sciences, Los Angeles, California

REFERENCES:
- [Derived] Wolitzky-Taylor K, Drazdowski TK, Niles A, Roy-Byrne P, Ries R, Rawson R, Craske MG. Change in anxiety sensitivity and substance use coping motives as putative mediators of treatment efficacy among substance users. Behav Res Ther. 2018 Aug;107:34-41. doi: 10.1016/j.brat.2018.05.010. Epub 2018 May 24. PMID 29852309
- [Derived] Wolitzky-Taylor K, Krull J, Rawson R, Roy-Byrne P, Ries R, Craske MG. Randomized clinical trial evaluating the preliminary effectiveness of an integrated anxiety disorder treatment in substance use disorder specialty clinics. J Consult Clin Psychol. 2018 Jan;86(1):81-88. doi: 10.1037/ccp0000276. PMID 29300100